CLINICAL TRIAL: NCT06526234
Title: Performance of Non-injected MR Enterography Compared to a Conventional MR Enterography Protocol With Contrast Agent Injection
Acronym: Fast-MR
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Valérie LAURENT, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2024PI153
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Crohn's disease or suspected Crohn's disease
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — MR enterography

SUMMARY:
Entero-MRI is indicated in Crohn's disease as part of the initial work-up or follow-up (to assess response to treatment, complications). The protocol for carrying out the examination complies with precise specifications set out in international recommendations. To perform the test, the small intestine must be distended with a hyperosmolar product. This protocol is applied to all patients, with no distinction or adaptation.

The total duration of the examination is sometimes difficult for patients to bear. Ingestion of the product to obtain distension of the small intestine is often poorly tolerated by patients.

In a number of cases, the entero-MRI may have been normal due to symptomatology regression or other diagnosis. The patient therefore underwent a complete examination similar to that of a patient with a pathology requiring characterization.

In this context, the investigators hypothesize that fast MR sequences are sufficient to discriminate between normal and abnormal examinations.

ELIGIBILITY:
Inclusion Criteria:

Patient with MR enterography examination for follow-up or suspected Crohn's disease

No Exclusion Criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with MR enterography examination for follow-up or suspected Crohn's disease
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Presence or absence of lesions detected visually by a radiologist on injection-free sequences versus conventional MR enterography. | Baseline (day 0)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, CHRU de Nancy, France